CLINICAL TRIAL: NCT05363319
Title: An Observational Study to Assess the Effectiveness and Safety of Cemiplimab Based Regimen in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) in Routine Clinical Practice Settings in Europe (CEMI-LUNG)
Brief Title: An Observational Study to Assess the Effectiveness and Safety of a Cemiplimab in Adult Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) in Routine Clinical Practice Settings in Europe
Acronym: CEMI-LUNG
Status: Recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R2810-ONC-2325; U1111-1275-9867 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab; Platinum Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Cemiplimab monotherapy
  Interventions: Drug: Cemiplimab
- Cohort 2: Cemiplimab in combination with platinum-based chemotherapy
  Interventions: Drug: Cemiplimab; Drug: Platinum-based chemotherapy

INTERVENTIONS:
Drug: Cemiplimab — solution for injection via intravenous (IV) infusion
  Other Names: SAR439684- Libtayo
Drug: Platinum-based chemotherapy — IV administration
  Groups: Cohort 2

SUMMARY:
This study is focused on patients with non-small cell lung cancer (NSCLC) and have been prescribed a cemiplimab (Libtayo®) based treatment regimen under standard care.

The goal of this study is to learn more about the use, benefits, and safety of cemiplimab based treatment regimens in participants with NSCLC.

DETAILED DESCRIPTION:
Originally registered as OBS17104 by Sanofi; transitioned to REGN 05Jul2023.

The recruitment period will be 48 months. Data will be collected during routine clinical visits approximately every three months while the patient is on cemiplimab treatment and then approximately every six months for up to 24 months after cemiplimab discontinuation. Patients will be followed from cemiplimab treatment initiation until death, loss to follow-up, study withdrawal, or to the end of the study period (72 months after study launch), whichever occurs first.

ELIGIBILITY:
Key Inclusion Criteria:

1. At least 18 years of age at the time of cemiplimab treatment initiation
2. Has been diagnosed with histologically or cytologically documented squamous or non-squamous NSCLC
3. Prescribed a cemiplimab-based regimen as part of routine clinical practice as determined by the treating physician per standard of care and in accordance with the Summary of Product Characteristics (SmPC).
4. Can understand and complete the study-related questionnaires
5. Must be legally capable of providing written consent for participation in the study and have signed informed consent prior to any study activities

Key Exclusion Criteria:

1. Has received cemiplimab prior to enrollment
2. Has uncontrolled autoimmune disease
3. Has a contraindication to cemiplimab as noted in the local SmPC
4. Is concurrently participating in any other study of an investigational drug or procedure
5. Has cognitive impairment or other medical condition that, in the opinion of the investigator, would interfere with the ability to complete the study-related questionnaires

NOTE: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this study will be patients with either locally advanced NSCLC not suitable for definitive chemoradiation or metastatic NSCLC and who are initiating a cemiplimab-based regimen of treatment as part of routine clinical practice at the time of study enrollment. The study will aim to enroll approximately 500 adult patients from up to 50 sites across Europe.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 72 months
  Date and primary cause of death

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 72 months
  Defined as the proportion of patients with a complete response or partial as the physician-reported best overall response.
Duration of Response (DoR) | Up to 72 months
  Defined among responders (patients with a complete response or partial response) as the time from the date of the first response after cemiplimab treatment initiation until the first date of disease progression or death due to any cause.
Time to Response (TTR) | Up to 72 months
  Defined as the time from the first cemiplimab dose until the date of first response observed for that patient. Patients who die during the study will be censored using the date of the last valid disease assessment).
Progression-Free Survival (PFS) | Up to 72 months
  Defined as the time from the first dose of cemiplimab until the date of the first documented tumour progression or death due to any cause.
Time to first subsequent anti-NSCLC treatment (TTST) | Up to 72 months
  Defined as the time from the first cemiplimab dose until the date of the first subsequent anti-NSCLC treatment.
Incidence of treatment-related adverse events (TR-AEs) in patients with advanced NSCLC treated with a cemiplimab-based regimen in routine clinical practice | Up to 72 months
  Number of patients with treatment related adverse events occurring during treatment
Incidence of treatment-related serious adverse events (TR-SAEs) in patients with advanced NSCLC treated with a cemiplimab-based regimen in routine clinical practice | Up to 72 months
  Number of patients with serious treatment related adverse events occurring during treatment
Incidence and severity of immune-mediated adverse events (imAEs) in patients with advanced NSCLC treated with a cemiplimab-based regimen in routine clinical practice | Up to 72 months
  Number of patients with immune-mediated adverse events and serious immune-mediated adverse events occurring during treatment
Incidence and severity of infusion related reactions (IRRs) in patients with advanced NSCLC treated with a cemiplimab-based regimen in routine clinical practice | Up to 72 months
  Number of patients with infusion related reactions and serious infusion related reactions adverse events occurring during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (48):
- Austria (2):
  - Klinikum Klagenfurt, Klagenfurt, Carinthia
  - Salzburger Landeskliniken (SALK), Salzburg, Salzburg
- France (9):
  - Le Groupe Hospitalier de la Region de Mulhouse et Sud Alsace, Emile Muller Hospital, Mulhouse, Alsace
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers, Nouvelle-Aquitaine
  - APHM - Hopital Nord, Marseille, Provenza
  - Hopitaux Universitaires de Strasbourg, Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire Angers, Angers
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - Center Hospitalier Universitaire (CHU) of Clermont, Clermont-Ferrand
  - Centre Hospitalier - Le mans, Le Mans
  - Hopital Tenon, Paris
- Germany (14):
  - Klinikum Konstanz, Konstanz, Baden-Wurttemberg
  - MedFISMO, Weinsberg, Baden-Wurttemberg
  - Staedtisches Klinikum Muenchen Bogenhausen, München, Bavaria
  - Franziskus Hospital Harderberg, Georgsmarienhütte, Georgsmarienhuette
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme), Großhansdorf, Schleswig-Holstein
  - St. Franziskus Hospital Münster, Münster, North Rhine-Westphalia
  - Haematologisch Onkologische Schwerpunktpraxis - Troisdorf, Troisdorf, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Gemeinschaftskrankenhaus Havelhoehe, Berlin
  - Gesellschaft fur Onkologische Studien Dortmund mbH (Gefos), Dortmund
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Pneumologische Praxis PD Dr. Med Christian Gessner, Leipzig
  - Marienhaus Klinikum Mainz, Mainz
  - Nuremberg Hospital, Campus North, Nuremberg
- Italy (12):
  - AO Universitaria Policlinico Vittorio Emanuele, Catania, Catania
  - Humanitas Istituto Clinico Catanese, Misterbianco, Catania
  - AOU Careggi, Florence, Firenze
  - IRCCS Humanitas Research Hospital, Rozzano, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena, Modena
  - AORN dei Colli, Napoli, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione G Pascale, Napoli, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - San Luigi Gonzaga University Hospital, Orbassano, Piedmont
  - Azienda Sanitaria Locale (ASL) Taranto, Taranto, Taranto
  - Ospedale Di Cisanello Azienda Ospedaliero Universitaria, Pisa, Tuscany
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
- Spain (11):
  - Hospital Torrecardenas, Almería, Almería
  - Hospital Universitario Virgen De La Victoria Malaga, Málaga, Andalusia
  - Parc Tauli Sabadell Hospital Universitari, Sabadell, Barcelona
  - Hospital Universitario De Jerez, Jerez de la Frontera, Cadiz
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
  - Complejo Hospitalario Universitario de Ferrol - Hospital Naval, Ferrol, Galicia
  - Hospital Universitario Alvaro Cunqueiro, Vigo, Pontevedra
  - University Hospital of Jaen, Jaén
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario Nuestra Senora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitari Sant Joan de Reus, Tarragona